CLINICAL TRIAL: NCT03631199
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study Evaluating the Efficacy and Safety of Pembrolizumab Plus Platinum-based Doublet Chemotherapy With or Without Canakinumab as First Line Therapy for Locally Advanced or Metastatic Non-squamous and Squamous Non-small Cell Lung Cancer Subjects (CANOPY-1)
Brief Title: Study of Efficacy and Safety of Pembrolizumab Plus Platinum-based Doublet Chemotherapy With or Without Canakinumab in Previously Untreated Locally Advanced or Metastatic Non-squamous and Squamous NSCLC Subjects
Acronym: CANOPY-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885U2301; 2024-511490-29-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ACZ885; canakinumab; pembrolizumab; carboplatin; cisplatin; paclitaxel; nab-paclitaxel; pemetrexed; NSCLC; non-small cell lung cancer; non small cell lung cancer; squamous; non-squamous; hsCRP; IL-1β; PD-L1; CANOPY; CANOPY-1; platinum-based doublet chemotherapy; first line therapy; locally advanced; metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — canakinumab; pembrolizumab; Carboplatin; Cisplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort A (Experimental): Safety run-in, canakinumab in combination with pembrolizumab, carboplatin, and pemetrexed.
  Interventions: Drug: canakinumab; Drug: pembrolizumab; Drug: carboplatin; Drug: pemetrexed
- Part 1: Cohort B (Experimental): Safety run-in, canakinumab in combination with pembrolizumab, cisplatin, and pemetrexed.
  Interventions: Drug: canakinumab; Drug: pembrolizumab; Drug: cisplatin; Drug: pemetrexed
- Part 1: Cohort C (Experimental): Safety run-in, canakinumab in combination with pembrolizumab, carboplatin, and paclitaxel.
  Interventions: Drug: canakinumab; Drug: pembrolizumab; Drug: carboplatin; Drug: paclitaxel
- Part 2: Canakinumab+pembro+CTx (Experimental): Double-blind, randomized, placebo-controlled, canakinumab in combination with pembrolizumab and platinum-based doublet chemotherapy.
  Interventions: Drug: canakinumab; Drug: pembrolizumab; Drug: carboplatin; Drug: cisplatin; Drug: paclitaxel; Drug: nab-paclitaxel; Drug: pemetrexed
- Part 2: Placebo+pembro+CTx (Other): Double-blind, randomized, placebo-controlled, canakinumab-matching placebo in combination with pembrolizumab and platinum-based doublet chemotherapy.
  Interventions: Drug: canakinumab-matching placebo; Drug: pembrolizumab; Drug: carboplatin; Drug: cisplatin; Drug: paclitaxel; Drug: nab-paclitaxel; Drug: pemetrexed

INTERVENTIONS:
Drug: canakinumab — canakinumab 200 mg subcutaneous (s.c.) injection every 3 weeks (squamous and non-squamous)
  Other Names: ACZ885
  Arms: Part 1: Cohort A; Part 1: Cohort B; Part 1: Cohort C; Part 2: Canakinumab+pembro+CTx
Drug: canakinumab-matching placebo — canakinumab placebo every 3 weeks (squamous and non-squamous)
  Arms: Part 2: Placebo+pembro+CTx
Drug: pembrolizumab — 200 mg every 3 weeks (squamous and non-squamous)
Drug: carboplatin — Area Under the Curve (AUC) 5 mg/mL*min every 3 weeks (non-squamous) or AUC 6 mg/mL*min (squamous)
  Arms: Part 1: Cohort A; Part 1: Cohort C; Part 2: Canakinumab+pembro+CTx; Part 2: Placebo+pembro+CTx
Drug: cisplatin — 75 mg/m^2 every 3 weeks (non-squamous)
  Arms: Part 1: Cohort B; Part 2: Canakinumab+pembro+CTx; Part 2: Placebo+pembro+CTx
Drug: paclitaxel — 200 mg/m^2 every 3 weeks (squamous)
  Arms: Part 1: Cohort C; Part 2: Canakinumab+pembro+CTx; Part 2: Placebo+pembro+CTx
Drug: nab-paclitaxel — 100 mg/m^2 on Days 1, 8, and 15 of every cycle (squamous)
  Arms: Part 2: Canakinumab+pembro+CTx; Part 2: Placebo+pembro+CTx
Drug: pemetrexed — 500 mg/m^2 every 3 weeks (non-squamous)
  Arms: Part 1: Cohort A; Part 1: Cohort B; Part 2: Canakinumab+pembro+CTx; Part 2: Placebo+pembro+CTx

SUMMARY:
This was a Phase III study of pembrolizumab plus platinum-based doublet chemotherapy with or without canakinumab in previously untreated locally advanced or metastatic non-squamous and squamous NSCLC participants.

DETAILED DESCRIPTION:
The study primarily assessed the safety and tolerability (safety run-in Part A) of pembrolizumab plus platinum-based doublet chemotherapy with canakinumab, and then, the efficacy (double-blind, randomized, placebo-controlled Part B) of pembrolizumab plus platinum-based doublet chemotherapy with or without canakinumab.

ELIGIBILITY:
Key inclusion criteria:

* Histologically confirmed locally advanced stage IIIB or stage IV NSCLC for treatment in the first-line setting
* Known PD-L1 status determined by a Novartis designated central laboratory. A newly obtained tissue biopsy or an archival biopsy (block or slides) is required for PD-L1 determination (PD-L1 IHC 22C3 pharmDx assay), prior to study randomization. Note: For the safety run-in part, known PD-L1 status is not required.
* Eastern Cooperative oncology group (ECOG) performance status of 0 or 1.
* At least 1 measurable lesion by RECIST 1.1

Key exclusion criteria:

* Previous immunotherapy (e.g. anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways).
* Prior treatment with canakinumab or drugs of a similar mechanism of action (IL-1β inhibitor).
* Subjects with epidermal growth factor receptor (EGFR) sensitizing mutations (identified in exons 19, 20, or 21), and/or ALK rearrangement by locally approved laboratory testing.
* Previously untreated or symptomatic central nervous system (CNS) metastases or lepto-meningeal disease.
* Subject with suspected or proven immune-compromised state or infections.
* Subject has prior to starting study drug: received live vaccination ≤3 months, had major surgery ≤4 weeks prior to starting study drug, has thoracic radiotherapy: lung fields ≤ 4 weeks, other anatomic sites ≤ 2 weeks, palliative radiotherapy for bone lesions ≤ 2 weeks.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2026-05-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (132):
- United States (4):
  - Pacific Shores Medical Group, Long Beach, California
  - USC Kenneth Norris Comprehensive Cancer Center, Los Angeles, California
  - AdventHealth, Orlando, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
- Argentina (2):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Caba
- Australia (4):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Austria (2):
  - Novartis Investigative Site, Linz, Upper Austria
  - Novartis Investigative Site, Salzburg
- Brazil (2):
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Chile (2):
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Santiago
- China (7):
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Valledupar, Cesar Department, Colombia
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Vitkovice
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Herning, Denmark
- Novartis Investigative Site, Oulu, Finland
- France (5):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (11):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Heidelberg
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Kowloon, Hong Kong
- Novartis Investigative Site, Veszprém, Hungary
- Novartis Investigative Site, Reykjavik, Iceland
- India (6):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Kolkata, West Bengal
- Italy (9):
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Orbassano, TO
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Ube, Yamaguchi
  - Novartis Investigative Site, Osaka
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Saida
- Malaysia (4):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Drammen, Norway
- Philippines (4):
  - Novartis Investigative Site, City of Taguig, National Capital Region
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Quezon
  - Novartis Investigative Site, San Juan City
- Poland (3):
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Tomaszw Mazowiecki
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (2):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Craiova, Dolj
- Russia (3):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Kosice-Saca
- South Korea (3):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (9):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Gipuzkoa
  - Novartis Investigative Site, Las Palmas de Gran C, Las Palmas
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Basel, Switzerland
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Bagcilar
  - Novartis Investigative Site, Ankara, Bilkent Cankaya
  - Novartis Investigative Site, Edirne, Merkez
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
- United Kingdom (4):
  - Novartis Investigative Site, High Heaton, Newcastle Upon Tyne
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Plymouth
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Tan DSW, Felip E, de Castro G, Solomon BJ, Greystoke A, Cho BC, Cobo M, Kim TM, Ganguly S, Carcereny E, Paz-Ares L, Bennouna J, Garassino MC, Schenker M, Kim SW, Brase JC, Bury-Maynard D, Passos VQ, Deudon S, Dharan B, Song Y, Caparica R, Johnson BE. Canakinumab Versus Placebo in Combination With First-Line Pembrolizumab Plus Chemotherapy for Advanced Non-Small-Cell Lung Cancer: Results From the CANOPY-1 Trial. J Clin Oncol. 2024 Jan 10;42(2):192-204. doi: 10.1200/JCO.23.00980. Epub 2023 Dec 1. PMID 38039427

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All inclusion and exclusion criteria were checked at screening.
Period: Overall Study
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Started | 10 | 11 | 9 | 320 | 323
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 11 | 9 | 320 | 323
Not completed — Progressive disease | 9 | 5 | 5 | 149 | 148
Not completed — Physician Decision | 0 | 2 | 3 | 19 | 13
Not completed — Adverse Event | 1 | 1 | 0 | 28 | 29
Not completed — Death | 0 | 1 | 0 | 35 | 48
Not completed — Subject decision | 0 | 1 | 0 | 12 | 12
Not completed — No treated | 0 | 0 | 0 | 0 | 1
Not completed — Treatment ongoing | 0 | 1 | 1 | 76 | 71
Not completed — Guardian decision | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx | Total
Number analyzed (Participants) | 10 | 11 | 9 | 320 | 323 | 673
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (6.57) | 57.9 (13.03) | 63.1 (7.18) | 61.7 (9.65) | 62.7 (8.74) | 62.2 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 3 | 93 | 91 | 192
  Male | 10 | 6 | 6 | 227 | 232 | 481
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 3 | 7 | 185 | 180 | 380
  Asian | 5 | 5 | 2 | 115 | 117 | 244
  Black or African American | 0 | 0 | 0 | 1 | 4 | 5
  Multiple | 0 | 0 | 0 | 0 | 2 | 2
  Missing | 0 | 3 | 0 | 19 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Part 1 (Safety Run-in): Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease progression, inter-current illness, or concomitant medications that met certain criteria as defined in the protocol.
Time Frame: During the first 42 days of dosing
Population: The dose-determining set (DDS) included all participants from the safety set who met the minimum exposure criterion and had sufficient safety evaluations, or experienced a dose-limiting toxicity (DLT) during the first 42 days (6 weeks) of dosing. Data are reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C
Number analyzed (Participants) | 10 | 10 | 9
Participants | 0 | 0 | 1

2. Primary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Progression-free Survival (PFS) Per Investigator Assessment Using RECIST v1.1
Description: Progression free survival was defined as the time from randomization to the date of the first documented radiological progression using RECIST 1.1 (Response evaluation criteria in solid tumor) or death due to any cause.
Time Frame: 18 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. Data are reported for Part 2 only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
months | 6.77 [5.62 to 7.75] | 6.77 [5.52 to 6.93]

3. Primary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Overall Survival (OS) Per Investigator Assessment Using RECIST v1.1
Description: Overall survival is defined as the time from date of randomization to date of death due to any cause.
Time Frame: Up to approximately 32 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
months | 20.83 [16.26 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 20.17 [16.23 to 22.37]

4. Secondary Outcome: Part 1 (Safety Run-in): Overall Response Rate (ORR) Per Investigator Assessment Using RECIST v1.1
Description: ORR was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR), as per investigator's assessment by RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 14 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. Data are reported for Part 1 only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C
Number analyzed (Participants) | 10 | 11 | 9
percentage of participants | 20.0 [2.5 to 55.6] | 72.7 [39.0 to 94.0] | 44.4 [13.7 to 78.8]

5. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Overall Response Rate (ORR) Per Investigator Assessment Using RECIST v1.1
Description: as for outcome 4
Time Frame: Up to approximately 26 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
percentage of participants | 45.6 [40.1 to 51.3] | 45.5 [40.0 to 51.1]

6. Secondary Outcome: Part 1 (Safety run-in): Disease Control Rate (DCR) Per Investigator Assessment Using RECIST v1.1
Description: Disease control rate was defined as the percentage of participants with complete response (CR) or partial response (PR) or participants with stable disease (SD) as per investigator assessment according to RECIST 1.1 criteria. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD=Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 14 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C
Number analyzed (Participants) | 10 | 11 | 9
percentage of participants | 70.0 [34.8 to 93.3] | 81.8 [48.2 to 97.7] | 77.8 [40.0 to 97.2]

7. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Disease Control Rate (DCR) Per Investigator Assessment Using RECIST v1.1
Description: as for outcome 6
Time Frame: Up to approximately 26 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
percentage of participants | 86.9 [82.7 to 90.4] | 84.8 [80.4 to 88.6]

8. Secondary Outcome: Part 1 (Safety run-in): Duration of Response (DOR) Per Investigator Assessment Using RECIST v1.1
Description: Duration of response was defined as the time from first documented response of CR or PR to date of first documented progression or death due to any cause, according to RECIST 1.1 criteria. DOR only applied to participants whose best overall response was CR or PR based on tumor response data per local review. If a participant did not have an event, DOR was censored at the date of last adequate tumor assessment. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 25 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. Participants who never achieved a best overall response of CR or PR were excluded from the analysis. Data are reported for responders in Part 1 only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C
Number analyzed (Participants) | 2 | 8 | 4
months | 7.43 [4.93 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 18.50 [6.34 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 8.15 [5.55 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

9. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Duration of Response (DOR) Per Investigator Assessment Using RECIST v1.1
Description: as for outcome 8
Time Frame: Up to approximately 26 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. Participants who never achieved a best overall response of CR or PR were excluded from the analysis. Data are reported for responders in Part 2 only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 146 | 147
months | 14.26 [10.41 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 13.60 [10.32 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

10. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Time to Response (TTR) Per Investigator Assessment Using RECIST v1.1
Description: Time to response (TTR) was defined as duration of time between the date of randomization and the date of first documented response of either CR or PR, according to RECIST 1.1 criteria. Duration of response was defined as the time from first documented response of CR or PR to date of first documented progression or death due to any cause, according to RECIST 1.1 criteria. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 26 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. Data are reported for responders in Part 2 only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 146 | 147
months | NA [8.94 to NA] — The median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [4.99 to NA] — The median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

11. Secondary Outcome: Part 1 (Safety Run-in): Antidrug Antibodies (ADA) of Canakinumab
Description: Participants with at least one ADA-positive sample.
Time Frame: Predose (0 hours (h)) on Day 1 of Cycles 1, 4, 8, 12, 16 (Cycle length =21 days), at end of treatment & then at 26, 78 and 130 days after last dose
Reporting Status: Not Posted, anticipated posting 2028-06

12. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Number of Participants With Antidrug Antibodies (ADA) of Canakinumab
Description: Participants with at least one ADA-positive sample.
Time Frame: Up to approximately 26 months
Population: The safety set comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. The data analysis applied to the Part 2 Canakinumab+pembro+CTx arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Canakinumab+Pembro+CTx
Number analyzed (Participants) | 320
Participants
  Baseline | 3
  On treatment | 2

13. Secondary Outcome: Part 1 (Safety run-in): Antidrug Antibodies (ADAs) of Pembrolizumab
Description: Participants with at least one ADA-positive sample.
Time Frame: Predose (0 h) on Day 1 of Cycles 1, 2, 4, 8, 12, 16 (Cycle length =21 days), at end of treatment & then at 26 days after last dose
Reporting Status: Not Posted, anticipated posting 2028-06

14. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Antidrug Antibodies (ADA) of Pembrolizumab
Description: Participants with at least one ADA-positive sample.
Time Frame: Up to approximately 26 months
Population: The safety set comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment. Data are reported for Part 2 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 322
Participants
  Baseline | 2 | 1
  On treatment | 7 | 2

15. Secondary Outcome: Part 1 (Safety Run-in): Serum Canakinumab Concentration
Time Frame: Predose (0 h) on Day 1 of Cycles 1-6, 8, 12, 16, Postdose on day 2, 8, 15 of Cycle 1, Post dose on Cycle 5 day 8, at end of treatment & then at 26, 78 and 130 days after last dose (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set - canakinumab included all participants who received at least one dose of canakinumab and had at least one evaluable PK sample for canakinumab. Data are reported for Part 1 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C
Number analyzed (Participants) | 9 | 11 | 9
μg/mL
  Cycle 1, Day 1, 0 hour n=9,11,9 | 0 (0) | 0 (0) | 0 (0)
  Cycle 1, Day 1, 24 hour n=8,11,9: number analyzed (Participants) | 8 | 11 | 9
  Cycle 1, Day 1, 24 hour n=8,11,9 | 4.43 (72.1) | 4.97 (113.5) | 4.57 (67.1)
  Cycle 1, Day 1, 168 hour n=9,11,9 | 12.1 (44.5) | 14.0 (61.7) | 12.8 (33.2)
  Cycle 1, Day 1, 336 hour n=8,10,8: number analyzed (Participants) | 8 | 10 | 8
  Cycle 1, Day 1, 336 hour n=8,10,8 | 11.1 (35.0) | 12.3 (55.2) | 10.9 (35.9)
  Cycle 2, Day 1, 0 hour n=9,9,7: number analyzed (Participants) | 9 | 9 | 7
  Cycle 2, Day 1, 0 hour n=9,9,7 | 10.2 (33.6) | 8.80 (49.4) | 8.69 (34.5)
  Cycle 3, Day 1, 0 hour n=7,9,8: number analyzed (Participants) | 7 | 9 | 8
  Cycle 3, Day 1, 0 hour n=7,9,8 | 16.9 (31.3) | 20.3 (40.3) | 17.1 (16.4)
  Cycle 4, Day 1, 0 hour n=8,8,6: number analyzed (Participants) | 8 | 8 | 6
  Cycle 4, Day 1, 0 hour n=8,8,6 | 23.1 (29.0) | 26.6 (35.0) | 19.4 (29.2)
  Cycle 5, Day 1, 0 hour n=4,7,6: number analyzed (Participants) | 4 | 7 | 6
  Cycle 5, Day 1, 0 hour n=4,7,6 | 26.9 (41.8) | 35.6 (47.6) | 22.4 (39.0)
  Cycle 5, Day 1, 168 hour n=5,9,4: number analyzed (Participants) | 5 | 9 | 4
  Cycle 5, Day 1, 168 hour n=5,9,4 | 32.1 (33.1) | 49.8 (42.5) | 32.7 (22.7)
  Cycle 6, Day 1, 0 hour n=3,7,6: number analyzed (Participants) | 3 | 7 | 6
  Cycle 6, Day 1, 0 hour n=3,7,6 | 32.2 (40.0) | 36.8 (47.8) | 26.3 (27.4)
  Cycle 8, Day 1, 0 hour n=3,7,4: number analyzed (Participants) | 3 | 7 | 4
  Cycle 8, Day 1, 0 hour n=3,7,4 | 37.7 (27.5) | 45.8 (38.6) | 29.9 (29.6)
  Cycle 12, Day 1, 0 hour n=2,6,4: number analyzed (Participants) | 2 | 6 | 4
  Cycle 12, Day 1, 0 hour n=2,6,4 | 40.6 (90.4) | 52.2 (42.9) | 32.4 (41.0)
  Cycle 16, Day 1, 0 hour n=1,5,4: number analyzed (Participants) | 1 | 5 | 4
  Cycle 16, Day 1, 0 hour n=1,5,4 | 68.2 (0) | 41.8 (67.3) | 31.0 (35.0)

16. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Serum Canakinumab Concentration
Time Frame: as for outcome 15
Population: The pharmacokinetic (PK) analysis set - canakinumab included all participants who received at least one dose of canakinumab and had at least one evaluable PK sample for canakinumab. Data are reported for the Part 2 Canakinumab+pembro+CTx arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx
Number analyzed (Participants) | 302
μg/mL
  Cycle 1, Day 1, 0 hour n=291: number analyzed (Participants) | 291
  Cycle 1, Day 1, 0 hour n=291 | 0 (0)
  Cycle 1, Day 1, 24 hour n=263: number analyzed (Participants) | 263
  Cycle 1, Day 1, 24 hour n=263 | 5.36 (99.3)
  Cycle 1, Day 1, 168 hour n=271: number analyzed (Participants) | 271
  Cycle 1, Day 1, 168 hour n=271 | 12.3 (52.1)
  Cycle 1, Day 1, 336 hour n=272: number analyzed (Participants) | 272
  Cycle 1, Day 1, 336 hour n=272 | 10.8 (47.2)
  Cycle 2, Day 1, 0 hour n=228: number analyzed (Participants) | 228
  Cycle 2, Day 1, 0 hour n=228 | 8.82 (46.8)
  Cycle 3, Day 1, 0 hour n=181: number analyzed (Participants) | 181
  Cycle 3, Day 1, 0 hour n=181 | 15.2 (40.1)
  Cycle 4, Day 1, 0 hour n=166: number analyzed (Participants) | 166
  Cycle 4, Day 1, 0 hour n=166 | 18.6 (44.4)
  Cycle 5, Day 1, 0 hour n=154: number analyzed (Participants) | 154
  Cycle 5, Day 1, 0 hour n=154 | 22.5 (42.9)
  Cycle 5, Day 1, 168 hour n=174: number analyzed (Participants) | 174
  Cycle 5, Day 1, 168 hour n=174 | 33.8 (42.2)
  Cycle 6, Day 1, 0 hour n=181: number analyzed (Participants) | 181
  Cycle 6, Day 1, 0 hour n=181 | 25.0 (47.5)
  Cycle 8, Day 1, 0 hour n=144: number analyzed (Participants) | 144
  Cycle 8, Day 1, 0 hour n=144 | 29.0 (46.9)
  Cycle 12, Day 1, 0 hour n=124: number analyzed (Participants) | 124
  Cycle 12, Day 1, 0 hour n=124 | 32.3 (49.8)
  Cycle 16, Day 1, 0 hour n=91: number analyzed (Participants) | 91
  Cycle 16, Day 1, 0 hour n=91 | 33.0 (49.0)

17. Secondary Outcome: Part 1 (Safety Run-in): Serum Pembrolizumab Concentration
Time Frame: Predose (0 h) on Day 1 of Cycles 1-6, 8, 12, 16, Postdose on day 2, 8, 15 of Cycle 1, at end of treatment & then at 26 days after last dose (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set -pembrolizumab included all participants who received at least one dose of pembrolizumab and had at least one evaluable PK sample for pembrolizumab. Data are reported for Part 1 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C
Number analyzed (Participants) | 9 | 11 | 9
μg/mL
  Cycle 1, Day 1, 0 hour n=9,11,9 | 0 (0) | 0 (0) | 0 (0)
  Cycle 1, Day 1, end-of-infusion, n=9,11,7: number analyzed (Participants) | 9 | 11 | 7
  Cycle 1, Day 1, end-of-infusion, n=9,11,7 | 53.9 (29.8) | 52.9 (41.9) | 48.1 (17.7)
  Cycle 1, Day 1, 24 hour n=7,11,9: number analyzed (Participants) | 7 | 11 | 9
  Cycle 1, Day 1, 24 hour n=7,11,9 | 40.5 (26.7) | 43.0 (35.1) | 41.4 (23.4)
  Cycle 1, Day 1, 168 hour n=9,11,9 | 19.0 (49.4) | 21.7 (42.9) | 18.7 (17.3)
  Cycle 1, Day 1, 336 hour n=9,11,8: number analyzed (Participants) | 9 | 11 | 8
  Cycle 1, Day 1, 336 hour n=9,11,8 | 15.1 (28.8) | 14.7 (40.6) | 12.5 (25.5)
  Cycle 2, Day 1, 0 hour n=9,9,7: number analyzed (Participants) | 9 | 9 | 7
  Cycle 2, Day 1, 0 hour n=9,9,7 | 12.2 (36.3) | 14.5 (49.2) | 10.5 (13.0)
  Cycle 3, Day 1, 0 hour n=7,9,7: number analyzed (Participants) | 7 | 9 | 7
  Cycle 3, Day 1, 0 hour n=7,9,7 | 21.0 (38.2) | 22.5 (46.8) | 15.5 (27.2)
  Cycle 4, Day 1, 0 hour n=8,8,6: number analyzed (Participants) | 8 | 8 | 6
  Cycle 4, Day 1, 0 hour n=8,8,6 | 27.8 (31.4) | 33.0 (108.5) | 23.5 (37.2)
  Cycle 5, Day 1, 0 hour n=5,7,6: number analyzed (Participants) | 5 | 7 | 6
  Cycle 5, Day 1, 0 hour n=5,7,6 | 28.6 (31.9) | 35.5 (44.3) | 28.5 (82.0)
  Cycle 5, Day 1, end-of-infusion n=5,7,5: number analyzed (Participants) | 5 | 7 | 5
  Cycle 5, Day 1, end-of-infusion n=5,7,5 | 77.7 (19.7) | 99.3 (29.6) | 57.4 (51.5)
  Cycle 6, Day 1, 0 hour n=2,7,5: number analyzed (Participants) | 2 | 7 | 5
  Cycle 6, Day 1, 0 hour n=2,7,5 | 30.6 (68.8) | 37.0 (33.6) | 26.6 (31.2)
  Cycle 8, Day 1, 0 hour n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Cycle 8, Day 1, 0 hour n=3,7,3 | 46.4 (16.2) | 45.3 (43.8) | 35.0 (52.0)
  Cycle 12, Day 1, 0 hour n=1,7,1: number analyzed (Participants) | 1 | 7 | 1
  Cycle 12, Day 1, 0 hour n=1,7,1 | 76.1 (0) | 42.9 (68.8) | 20.5 (0)
  Cycle 16, Day 1, 0 hour n=1,5,1: number analyzed (Participants) | 1 | 5 | 1
  Cycle 16, Day 1, 0 hour n=1,5,1 | 39.8 (0) | 43.4 (84.5) | 27.2 (0)

18. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Serum Pembrolizumab Concentration
Time Frame: as for outcome 17
Population: The pharmacokinetic (PK) analysis set -pembrolizumab included all participants who received at least one dose of pembrolizumab and had at least one evaluable PK sample for pembrolizumab. Data are reported for Part 2 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 36 | 36
μg/mL
  Cycle 1, Day 1, 0 hours n=29,28: number analyzed (Participants) | 29 | 28
  Cycle 1, Day 1, 0 hours n=29,28 | 0 (0) | 0 (0)
  Cycle 1, Day 1, end-of-infusion, n=27,27: number analyzed (Participants) | 27 | 27
  Cycle 1, Day 1, end-of-infusion, n=27,27 | 53.5 (55.1) | 50.9 (36.0)
  Cycle 1, Day 1, 24 hours n=29,31: number analyzed (Participants) | 29 | 31
  Cycle 1, Day 1, 24 hours n=29,31 | 45.9 (23.6) | 43.7 (51.8)
  Cycle 1, Day 1, 168 hours n=28,29: number analyzed (Participants) | 28 | 29
  Cycle 1, Day 1, 168 hours n=28,29 | 21.5 (30.1) | 21.4 (42.2)
  Cycle 1, Day 1, 336 hours n=23,25: number analyzed (Participants) | 23 | 25
  Cycle 1, Day 1, 336 hours n=23,25 | 14.5 (33.8) | 14.9 (39.9)
  Cycle 2, Day 1, 0 hours n=19,25: number analyzed (Participants) | 19 | 25
  Cycle 2, Day 1, 0 hours n=19,25 | 11.5 (46.6) | 12.9 (39.3)
  Cycle 3, Day 1, 0 hours n=12,20: number analyzed (Participants) | 12 | 20
  Cycle 3, Day 1, 0 hours n=12,20 | 22.7 (39.8) | 20.6 (50.0)
  Cycle 4, Day 1, 0 hours n=12,20: number analyzed (Participants) | 12 | 20
  Cycle 4, Day 1, 0 hours n=12,20 | 24.7 (42.5) | 27.2 (55.0)
  Cycle 5, Day 1, 0 hours n=15,22: number analyzed (Participants) | 15 | 22
  Cycle 5, Day 1, 0 hours n=15,22 | 28.6 (38.6) | 26.5 (55.0)
  Cycle 5, Day 1, end-of-infusion n=18,21: number analyzed (Participants) | 18 | 21
  Cycle 5, Day 1, end-of-infusion n=18,21 | 66.3 (42.6) | 70.9 (41.5)
  Cycle 6, Day 1, 0 hours n=14,17: number analyzed (Participants) | 14 | 17
  Cycle 6, Day 1, 0 hours n=14,17 | 34.0 (69.0) | 32.2 (71.5)
  Cycle 8, Day 1, 0 hours n=16,17: number analyzed (Participants) | 16 | 17
  Cycle 8, Day 1, 0 hours n=16,17 | 36.0 (53.2) | 30.1 (57.4)
  Cycle 12, Day 1, 0 hours n=10,9: number analyzed (Participants) | 10 | 9
  Cycle 12, Day 1, 0 hours n=10,9 | 47.6 (27.6) | 41.9 (44.7)
  Cycle 16, Day 1, 0 hours n=9,8: number analyzed (Participants) | 9 | 8
  Cycle 16, Day 1, 0 hours n=9,8 | 42.9 (39.4) | 47.0 (38.0)

19. Secondary Outcome: Part 1 (Safety Run-in): Plasma Pemetrexed Concentration
Time Frame: Predose (0 h) and end of infusion on Cycle 1 and 2; 1, 4, 8 h post infusion on Cycle 1; 1, 2, 4, 8h post infusion on Cycle 2 (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set -pemetrexed included all participants who received at least one dose of pemetrexed and had at least one evaluable PK sample for pemetrexed. Data are reported for the Part 1 Cohorts A and B arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort A | Part 1: Cohort B
Number analyzed (Participants) | 9 | 11
μg/mL
  Cycle 1, Day 1, Pre-infusion n=9,11 | 0 (0) | 517 (1.4)
  Cycle 1, Day 1, end-of-infusion, n=9,11 | 102000 (30.2) | 87800 (39.5)
  Cycle 1, Day 1, 1 hour n=9,11 | 39000 (23.3) | 39000 (29.5)
  Cycle 1, Day 1, 4 hours n=9,11 | 10300 (25.1) | 10300 (29.6)
  Cycle 1, Day 1, 8 hours n=9,11 | 3180 (38.3) | 2340 (58.8)
  Cycle 2, Day 1, Pre-infusion n=8,10: number analyzed (Participants) | 8 | 10
  Cycle 2, Day 1, Pre-infusion n=8,10 | 0 (0) | 0 (0)
  Cycle 2, Day 1, End-of-infusion n=9,10: number analyzed (Participants) | 9 | 10
  Cycle 2, Day 1, End-of-infusion n=9,10 | 93300 (19.0) | 92600 (37.5)
  Cycle 2, Day 1, 1 hour n=9,10: number analyzed (Participants) | 9 | 10
  Cycle 2, Day 1, 1 hour n=9,10 | 43600 (15.7) | 43500 (16.2)
  Cycle 2, Day 1, 2 hours n=9,9: number analyzed (Participants) | 9 | 9
  Cycle 2, Day 1, 2 hours n=9,9 | 26300 (19.1) | 23400 (13.9)
  Cycle 2, Day 1, 4 hours n=9,10: number analyzed (Participants) | 9 | 10
  Cycle 2, Day 1, 4 hours n=9,10 | 11100 (25.5) | 10800 (34.3)
  Cycle 2, Day 1, 8 hours n=9,10: number analyzed (Participants) | 9 | 10
  Cycle 2, Day 1, 8 hours n=9,10 | 3920 (39.1) | 2760 (55.0)

20. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Plasma Pemetrexed Concentration
Time Frame: as for outcome 19
Population: The pharmacokinetic (PK) analysis set -pemetrexed included all participants who received at least one dose of pemetrexed and had at least one evaluable PK sample for pemetrexed. Data are reported for Part 2 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 19 | 20
μg/mL
  Cycle 1, Day 1, Pre-infusion n=18,18: number analyzed (Participants) | 18 | 18
  Cycle 1, Day 1, Pre-infusion n=18,18 | 0 (0) | 0 (0)
  Cycle 1, Day 1, end-of-infusion, n=19,20 | 92000 (21.9) | 86400 (46.6)
  Cycle 1, Day 1, 1 hour n=19,20 | 42900 (23.5) | 36900 (29.4)
  Cycle 1, Day 1, 4 hours n=19,20 | 11700 (33.3) | 9390 (48.5)
  Cycle 2, Day 1, Pre-infusion n=15,16: number analyzed (Participants) | 15 | 16
  Cycle 2, Day 1, Pre-infusion n=15,16 | 0 (0) | 0 (0)
  Cycle 2, Day 1, End-of-infusion n=15,17: number analyzed (Participants) | 15 | 17
  Cycle 2, Day 1, End-of-infusion n=15,17 | 89200 (40.8) | 97000 (32.3)
  Cycle 2, Day 1, 1 hour n=15,17: number analyzed (Participants) | 15 | 17
  Cycle 2, Day 1, 1 hour n=15,17 | 47600 (30.9) | 37300 (20.6)
  Cycle 2, Day 1, 2 hours n=15,17: number analyzed (Participants) | 15 | 17
  Cycle 2, Day 1, 2 hours n=15,17 | 26900 (28.7) | 20900 (41.9)
  Cycle 2, Day 1, 4 hours n=14,17: number analyzed (Participants) | 14 | 17
  Cycle 2, Day 1, 4 hours n=14,17 | 12500 (38.2) | 9880 (55.8)

21. Secondary Outcome: Part 1 (Safety Run-in): Plasma Cisplatin Concentration
Time Frame: Predose (0 h) and end of infusion on Cycle 1 and 2; 2, 4, 8 h post infusion on Cycle 1; 1.5, 2, 4, 8 h post infusion on Cycle 2 (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set -cisplatin included all participants who received at least one dose of cisplatin and had at least one evaluable PK sample for cisplatin. Data are reported for the Part 1 Cohort B arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort B
Number analyzed (Participants) | 11
μg/mL
  Cycle 1, Day 1, Pre-infusion n=11 | 0 (0)
  Cycle 1, Day 1, end-of-infusion, n=11 | 3750 (130.2)
  Cycle 1, Day 1, 2 hours n=6: number analyzed (Participants) | 6
  Cycle 1, Day 1, 2 hours n=6 | 3690 (248.2)
  Cycle 1, Day 1, 4 hours n=11 | 1930 (35.9)
  Cycle 1, Day 1, 8 hours n=11 | 1680 (22.4)
  Cycle 2, Day 1, Pre-infusion n=10: number analyzed (Participants) | 10
  Cycle 2, Day 1, Pre-infusion n=10 | 235 (29.3)
  Cycle 2, Day 1, End-of-infusion n=10: number analyzed (Participants) | 10
  Cycle 2, Day 1, End-of-infusion n=10 | 2900 (45.6)
  Cycle 2, Day 1, 1.5 hours n=10: number analyzed (Participants) | 10
  Cycle 2, Day 1, 1.5 hours n=10 | 2100 (51.9)
  Cycle 2, Day 1, 2 hours n=5: number analyzed (Participants) | 5
  Cycle 2, Day 1, 2 hours n=5 | 2650 (20.3)
  Cycle 2, Day 1, 4 hours n=10: number analyzed (Participants) | 10
  Cycle 2, Day 1, 4 hours n=10 | 2070 (15.2)
  Cycle 2, Day 1, 8 hours n=10: number analyzed (Participants) | 10
  Cycle 2, Day 1, 8 hours n=10 | 1750 (29.9)

22. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Plasma Cisplatin Concentration
Time Frame: Predose (0 h) and end of infusion on Cycle 1 and 2; 2, 4, 8 h post infusion on Cycle 1; 1.5, 2, 4, 8 h post infusion on Cycle 2 (Cycle length = 21 days)
Population: The pharmacokinetic (PK) analysis set -cisplatin included all participants who received at least one dose of cisplatin and had at least one evaluable PK sample for cisplatin. Data are reported for Part 2 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 23 | 19
μg/mL
  Cycle 1, Day 1, Pre-infusion n=21,18: number analyzed (Participants) | 21 | 18
  Cycle 1, Day 1, Pre-infusion n=21,18 | 0 (0) | 177 (47.5)
  Cycle 1, Day 1, end-of-infusion, n=20,18: number analyzed (Participants) | 20 | 18
  Cycle 1, Day 1, end-of-infusion, n=20,18 | 3670 (49.6) | 3120 (20.9)
  Cycle 1, Day 1, 2 hours n=17,18: number analyzed (Participants) | 17 | 18
  Cycle 1, Day 1, 2 hours n=17,18 | 2280 (27.8) | 2180 (23.5)
  Cycle 1, Day 1, 4 hours n=17,16: number analyzed (Participants) | 17 | 16
  Cycle 1, Day 1, 4 hours n=17,16 | 1950 (11.2) | 1950 (17.5)
  Cycle 2, Day 1, Pre-infusion n=20,14: number analyzed (Participants) | 20 | 14
  Cycle 2, Day 1, Pre-infusion n=20,14 | 288 (58.9) | 296 (51.7)
  Cycle 2, Day 1, End-of-infusion n=19,13: number analyzed (Participants) | 19 | 13
  Cycle 2, Day 1, End-of-infusion n=19,13 | 3130 (92.0) | 2820 (88.2)
  Cycle 2, Day 1, 1.5 hours n=16,12: number analyzed (Participants) | 16 | 12
  Cycle 2, Day 1, 1.5 hours n=16,12 | 2790 (29.9) | 2410 (38.3)
  Cycle 2, Day 1, 2 hours n=16,12: number analyzed (Participants) | 16 | 12
  Cycle 2, Day 1, 2 hours n=16,12 | 2550 (22.7) | 2790 (23.9)
  Cycle 2, Day 1, 4 hours n=19,11: number analyzed (Participants) | 19 | 11
  Cycle 2, Day 1, 4 hours n=19,11 | 2340 (17.4) | 2340 (13.7)

23. Secondary Outcome: Part 1 (Safety Run-in): Plasma Carboplatin Concentration
Time Frame: Predose (0 h), end of infusion, 1, 2, 4, 8 h post infusion on Cycles 1 and 2 (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set -carboplatin included all participants who received at least one dose of carboplatin and had at least one evaluable PK sample for carboplatin. Data are reported for the Part 1 Cohorts A and C arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort A | Part 1: Cohort C
Number analyzed (Participants) | 9 | 9
μg/mL
  Cycle 1, Day 1, Pre-infusion n=8,9: number analyzed (Participants) | 8 | 9
  Cycle 1, Day 1, Pre-infusion n=8,9 | 0 (0) | 0 (0)
  Cycle 1, Day 1, End-of-infusion, n=9,9 | 17400 (21.9) | 21700 (49.8)
  Cycle 1, Day 1, 1 hour n=9,6: number analyzed (Participants) | 9 | 6
  Cycle 1, Day 1, 1 hour n=9,6 | 10400 (42.7) | 13300 (46.8)
  Cycle 1, Day 1, 2 hours n=9,9 | 6200 (34.3) | 7380 (23.5)
  Cycle 1, Day 1, 4 hours n=9,9 | 3380 (34.6) | 3970 (29.4)
  Cycle 1, Day 1, 8 hours n=9,6: number analyzed (Participants) | 9 | 6
  Cycle 1, Day 1, 8 hours n=9,6 | 1370 (33.6) | 1540 (39.6)
  Cycle 2, Day 1, Pre-infusion n=9,9 | 125 (29.7) | 120 (16.4)
  Cycle 2, Day 1, End-of-infusion n=9,9 | 10300 (441.8) | 16200 (32.4)
  Cycle 2, Day 1, 1 hour n=8,6: number analyzed (Participants) | 8 | 6
  Cycle 2, Day 1, 1 hour n=8,6 | 13300 (44.1) | 11400 (24.5)
  Cycle 2, Day 1, 2 hours n=9,9 | 8080 (38.5) | 6620 (22.5)
  Cycle 2, Day 1, 4 hours n=9,9 | 3590 (26.8) | 3680 (26.7)
  Cycle 2, Day 1, 8 hours n=9,5: number analyzed (Participants) | 9 | 5
  Cycle 2, Day 1, 8 hours n=9,5 | 1670 (29.7) | 1800 (34.8)

24. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Plasma Carboplatin Concentration
Time Frame: Predose (0 h), end of infusion, 1, 2, 4, 8 h post infusion on Cycles 1 and 2 (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set -carboplatin included all participants who received at least one dose of carboplatin and had at least one evaluable PK sample for carboplatin. Data are reported for Part 2 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 18 | 23
μg/mL
  Cycle 1, Day 1, Pre-infusion n=17,19: number analyzed (Participants) | 17 | 19
  Cycle 1, Day 1, Pre-infusion n=17,19 | 0 (0) | 668 (0)
  Cycle 1, Day 1, End-of-infusion, n=17,23: number analyzed (Participants) | 17 | 23
  Cycle 1, Day 1, End-of-infusion, n=17,23 | 13800 (23.4) | 16900 (53.6)
  Cycle 1, Day 1, 1 hour n=14,21: number analyzed (Participants) | 14 | 21
  Cycle 1, Day 1, 1 hour n=14,21 | 9980 (40.4) | 10600 (35.9)
  Cycle 1, Day 1, 2 hours n=17,23: number analyzed (Participants) | 17 | 23
  Cycle 1, Day 1, 2 hours n=17,23 | 7250 (25.0) | 6930 (36.3)
  Cycle 1, Day 1, 4 hours n=16,22: number analyzed (Participants) | 16 | 22
  Cycle 1, Day 1, 4 hours n=16,22 | 3690 (26.4) | 3780 (46.7)
  Cycle 2, Day 1, Pre-infusion n=11,16: number analyzed (Participants) | 11 | 16
  Cycle 2, Day 1, Pre-infusion n=11,16 | 145 (37.2) | 121 (8.6)
  Cycle 2, Day 1, End-of-infusion n=11,18: number analyzed (Participants) | 11 | 18
  Cycle 2, Day 1, End-of-infusion n=11,18 | 14300 (34.8) | 13000 (183.5)
  Cycle 2, Day 1, 1 hour n=10,16: number analyzed (Participants) | 10 | 16
  Cycle 2, Day 1, 1 hour n=10,16 | 8880 (23.8) | 9490 (213.7)
  Cycle 2, Day 1, 2 hours n=12,18: number analyzed (Participants) | 12 | 18
  Cycle 2, Day 1, 2 hours n=12,18 | 6810 (35.3) | 7080 (26.5)
  Cycle 2, Day 1, 4 hours n=11,18: number analyzed (Participants) | 11 | 18
  Cycle 2, Day 1, 4 hours n=11,18 | 3990 (34.4) | 3830 (37.4)

25. Secondary Outcome: Part 1 (Safety Run-in): Plasma Paclitaxel Concentration
Time Frame: Predose (0 h) and end of infusion on Cycle 1 and 2; 4, 8, 12 h post infusion on Cycle 1; 4, 6, 8, 12 h post infusion on Cycle 2 (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set -paclitaxel included all participants who received at least one dose of paclitaxel and had at least one evaluable PK sample for paclitaxel. Data are reported for the Part 1 Cohort C arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort C
Number analyzed (Participants) | 9
μg/mL
  Cycle 1, Day 1, Pre-infusion n=9 | 0 (0)
  Cycle 1, Day 1, End-of-infusion, n=9 | 4440 (42.5)
  Cycle 1, Day 1, 4 hours n=8: number analyzed (Participants) | 8
  Cycle 1, Day 1, 4 hours n=8 | 827 (111.3)
  Cycle 1, Day 1, 8 hours n=9 | 310 (83.5)
  Cycle 1, Day 1, 12 hours n=6: number analyzed (Participants) | 6
  Cycle 1, Day 1, 12 hours n=6 | 130 (78.3)
  Cycle 2, Day 1, Pre-infusion n=7: number analyzed (Participants) | 7
  Cycle 2, Day 1, Pre-infusion n=7 | 0 (0)
  Cycle 2, Day 1, End-of-infusion n=7: number analyzed (Participants) | 7
  Cycle 2, Day 1, End-of-infusion n=7 | 4940 (35.1)
  Cycle 2, Day 1, 4 hours n=7: number analyzed (Participants) | 7
  Cycle 2, Day 1, 4 hours n=7 | 1090 (89.5)
  Cycle 2, Day 1, 6 hours n=8: number analyzed (Participants) | 8
  Cycle 2, Day 1, 6 hours n=8 | 525 (74.1)
  Cycle 2, Day 1, 8 hours n=7: number analyzed (Participants) | 7
  Cycle 2, Day 1, 8 hours n=7 | 333 (79.8)
  Cycle 2, Day 1, 12 hours n=4: number analyzed (Participants) | 4
  Cycle 2, Day 1, 12 hours n=4 | 134 (89.7)

26. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Plasma Paclitaxel Concentration
Time Frame: as for outcome 25
Population: The pharmacokinetic (PK) analysis set -paclitaxel included all participants who received at least one dose of paclitaxel and had at least one evaluable PK sample for paclitaxel. Data are reported for Part 2 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 14 | 13
μg/mL
  Cycle 1, Day 1, Pre-infusion n=12,11: number analyzed (Participants) | 12 | 11
  Cycle 1, Day 1, Pre-infusion n=12,11 | 0 (0) | 0 (0)
  Cycle 1, Day 1, End-of-infusion, n=13,12: number analyzed (Participants) | 13 | 12
  Cycle 1, Day 1, End-of-infusion, n=13,12 | 4620 (97.3) | 3380 (116.8)
  Cycle 1, Day 1, 4 hours n=12,11: number analyzed (Participants) | 12 | 11
  Cycle 1, Day 1, 4 hours n=12,11 | 1880 (43.5) | 1900 (88.4)
  Cycle 1, Day 1, 24 hours n=10,8: number analyzed (Participants) | 10 | 8
  Cycle 1, Day 1, 24 hours n=10,8 | 102 (38.9) | 114 (47.4)
  Cycle 2, Day 1, Pre-infusion n=9,8: number analyzed (Participants) | 9 | 8
  Cycle 2, Day 1, Pre-infusion n=9,8 | 0 (0) | 0 (0)
  Cycle 2, Day 1, End-of-infusion n=10,9: number analyzed (Participants) | 10 | 9
  Cycle 2, Day 1, End-of-infusion n=10,9 | 3930 (41.8) | 3660 (75.1)
  Cycle 2, Day 1, 4 hours n=9,9: number analyzed (Participants) | 9 | 9
  Cycle 2, Day 1, 4 hours n=9,9 | 1450 (26.6) | 1180 (62.6)
  Cycle 2, Day 1, 6 hours n=7,8: number analyzed (Participants) | 7 | 8
  Cycle 2, Day 1, 6 hours n=7,8 | 920 (45.7) | 775 (55.0)
  Cycle 2, Day 1, 24 hours n=10,7: number analyzed (Participants) | 10 | 7
  Cycle 2, Day 1, 24 hours n=10,7 | 101 (23.6) | 81.4 (27.7)

27. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Plasma Nab-paclitaxel Concentration
Time Frame: Predose (0 h) and end of infusion on Cy 1 and 2, 4, 8, 12 h post infusion on Cy 1, 4, 6, 8, 12 h post infusion on Cy 2 (Cy length =21 days)
Population: The pharmacokinetic (PK) analysis set -nab-paclitaxel included all participants who received at least one dose of nab-paclitaxel and had at least one evaluable PK sample for nab-paclitaxel. Data are reported for Part 2 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 11 | 15
μg/mL
  Cycle 1, Day 1, Pre-infusion n=9,13: number analyzed (Participants) | 9 | 13
  Cycle 1, Day 1, Pre-infusion n=9,13 | 0 (0) | 0 (0)
  Cycle 1, Day 1, End-of-infusion, n=10,15: number analyzed (Participants) | 10 | 15
  Cycle 1, Day 1, End-of-infusion, n=10,15 | 2620 (87.5) | 2520 (285.4)
  Cycle 1, Day 1, 4 hours n=10,14: number analyzed (Participants) | 10 | 14
  Cycle 1, Day 1, 4 hours n=10,14 | 112 (38.3) | 117 (90.2)
  Cycle 1, Day 1, 24 hours n=4,9: number analyzed (Participants) | 4 | 9
  Cycle 1, Day 1, 24 hours n=4,9 | 24.2 (16.7) | 23.9 (47.8)
  Cycle 2, Day 1, Pre-infusion n=7,8: number analyzed (Participants) | 7 | 8
  Cycle 2, Day 1, Pre-infusion n=7,8 | 0 (0) | 44.6 (160.1)
  Cycle 2, Day 1, End-of-infusion n=7,8: number analyzed (Participants) | 7 | 8
  Cycle 2, Day 1, End-of-infusion n=7,8 | 1630 (92.1) | 3440 (79.1)
  Cycle 2, Day 1, 4 hours n=6,8: number analyzed (Participants) | 6 | 8
  Cycle 2, Day 1, 4 hours n=6,8 | 83.6 (45.5) | 96.5 (63.8)
  Cycle 2, Day 1, 6 hours n=6,8: number analyzed (Participants) | 6 | 8
  Cycle 2, Day 1, 6 hours n=6,8 | 75.6 (47.1) | 86.1 (55.2)
  Cycle 2, Day 1, 24 hours n=5,7: number analyzed (Participants) | 5 | 7
  Cycle 2, Day 1, 24 hours n=5,7 | 34.5 (107.7) | 23.6 (39.2)

28. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Time to Definitive 10-point Deterioration (TTDD) Symptom Scores of Pain, Cough and Dyspnea Per EORTC QLQ-LC13 Questionnaire
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, dyspnea, and chest pain). Scores for each scale and single-item range from 0 to 100, with higher scores indicating higher level of symptoms. TTDD for chest pain, cough and dyspnea was defined as the time from randomization to the date of event, which was defined as at least 10 points absolute worsening from baseline of the corresponding scale score, with no later change below this threshold ie.<10 points was observed, or if this worsening was observed at the last assessment for the subject, or death due to any cause (whichever occurred earlier). If a subject did not have an event, TTDD was censored at the last adequate assessment.
Time Frame: Up to approximately 25 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
months
  Chest Pain n=65,96: number analyzed (Participants) | 65 | 96
  Chest Pain n=65,96 | NA [NA to NA] — The median and lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | 22.14 [18.40 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
  Cough n=63,94: number analyzed (Participants) | 63 | 94
  Cough n=63,94 | NA [NA to NA] — The median and lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | 23.06 [17.51 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
  Dyspnea n=111,149: number analyzed (Participants) | 111 | 149
  Dyspnea n=111,149 | 19.61 [13.50 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 11.50 [7.66 to 15.90]
Statistical Analysis 1: Comparison: Part 2: Canakinumab+Pembro+CTx vs Part 2: Placebo+Pembro+CTx; Chest pain; Test type: Equivalence — Nominal p-values are presented without any statistical inference since there was no adjustment for multiplicity; p = 0.00164, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.45 to 0.86]
Statistical Analysis 2: Comparison: Part 2: Canakinumab+Pembro+CTx vs Part 2: Placebo+Pembro+CTx; Cough; Test type: Equivalence — Nominal p-values are presented without any statistical inference since there was no adjustment for multiplicity; p = 0.00069, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.43 to 0.82]
Statistical Analysis 3: Comparison: Part 2: Canakinumab+Pembro+CTx vs Part 2: Placebo+Pembro+CTx; Dyspnea; Test type: Equivalence — Nominal p-values are presented without any statistical inference since there was no adjustment for multiplicity; p = 0.00045, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.51 to 0.84]

29. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Time to Definitive Deterioration in Global Health Status/Quality of Life, Shortness of Breath and Pain Per EORTC QLQ-C30 Questionnaire
Description: The European Organization for Research and Treatment of Cancer quality of life (EORTC QLQ-C30) is a questionnaire developed to assess the health-related quality of life of cancer participants. It assesses 15 domains consisting of 5 functional domains (physical, role, emotional, cognitive, social) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global health status/QoL scale. All domain scores range from 0 to 100. A high score for the functional or global health status scales indicates a high level of functioning or QoL; a high score for a symptom scale indicates a high level of symptoms.
Time Frame: Up to approximately 25 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
months
  Quality of Life n=119, 129: number analyzed (Participants) | 119 | 129
  Quality of Life n=119, 129 | 17.54 [14.06 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 15.90 [11.40 to 20.04]
  Shortness of Breath n=83,115: number analyzed (Participants) | 83 | 115
  Shortness of Breath n=83,115 | NA [NA to NA] — The median and lower and upper limits of 95% CI were not estimable due to an insufficient number of participants with events. | 19.29 [14.13 to 21.62]
  Pain n=117,122: number analyzed (Participants) | 117 | 122
  Pain n=117,122 | 20.07 [13.24 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 17.91 [12.65 to 22.11]
Statistical Analysis 1: Comparison: Part 2: Canakinumab+Pembro+CTx vs Part 2: Placebo+Pembro+CTx; Quality of Life; Test type: Equivalence — Nominal p-values are presented without any statistical inference since there was no adjustment for multiplicity; p = 0.113, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.66 to 1.10]
Statistical Analysis 2: Comparison: Part 2: Canakinumab+Pembro+CTx vs Part 2: Placebo+Pembro+CTx; Shortness of Breath; Test type: Equivalence — Nominal p-values are presented without any statistical inference since there was no adjustment for multiplicity; p = 0.00433, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.51 to 0.91]
Statistical Analysis 3: Comparison: Part 2: Canakinumab+Pembro+CTx vs Part 2: Placebo+Pembro+CTx; Pain; Test type: Equivalence — Nominal p-values are presented without any statistical inference since there was no adjustment for multiplicity; p = 0.294, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.72 to 1.20]

30. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Change From Baseline in Score as Per the EuroQol 5 Dimension 5 Level (EQ-5D-5L) Questionnaire
Description: The EQ-5D-5L questionnaire is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L measures 5 items on mobility, self-care, usual activities, pain/discomfort, anxiety/depression, measured on 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A utility index can be computed from the EQ 5D-5L descriptive system with utility scores ranging from -0.281 (worst imaginable health state) to 1 (best imaginable health state), with -0.281 representing an "unconscious" health state. A single index value is analyzed for the EQ-5D-5L score. An increase from baseline in the EQ-ED-5L utility index is indicative of an improvement.). CFB = change from baseline
Time Frame: Assessed every 3 weeks from Week 3 through Week 108, at follow-up visits 1, 2, 3, 4, and 5 (follow-up visits occurred every 26 days from week 108), and at 7 and 28 days post-disease progression, all up to a maximum of 3.5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
score on a scale
  CFB at Week 3 n=254,249: number analyzed (Participants) | 254 | 249
  CFB at Week 3 n=254,249 | 0.766 (0.2138) | 0.768 (0.2153)
  CFB at Week 6 n=236,230: number analyzed (Participants) | 236 | 230
  CFB at Week 6 n=236,230 | 0.029 (0.2135) | 0.032 (0.2317)
  CFB at Week 9 n=220,219: number analyzed (Participants) | 220 | 219
  CFB at Week 9 n=220,219 | 0.019 (0.2074) | 0.059 (0.2512)
  CFB at Week 12 n=192,214: number analyzed (Participants) | 192 | 214
  CFB at Week 12 n=192,214 | 0.028 (0.2101) | 0.044 (0.2486)
  CFB at Week 15 n=194,196: number analyzed (Participants) | 194 | 196
  CFB at Week 15 n=194,196 | 0.031 (0.2103) | 0.039 (0.2512)
  CFB at Week 18 n=187,198: number analyzed (Participants) | 187 | 198
  CFB at Week 18 n=187,198 | 0.020 (0.2192) | 0.050 (0.2723)
  CFB at Week 21 n=173,176: number analyzed (Participants) | 173 | 176
  CFB at Week 21 n=173,176 | 0.016 (0.2291) | 0.041 (0.2533)
  CFB at Week 24 n=160,164: number analyzed (Participants) | 160 | 164
  CFB at Week 24 n=160,164 | 0.027 (0.2062) | 0.050 (0.2824)
  CFB at Week 27 n=157,155: number analyzed (Participants) | 157 | 155
  CFB at Week 27 n=157,155 | 0.020 (0.1929) | 0.043 (0.2828)
  CFB at Week 30 n=140,145: number analyzed (Participants) | 140 | 145
  CFB at Week 30 n=140,145 | 0.047 (0.1928) | 0.046 (0.2897)
  CFB at Week 33 n=136,124: number analyzed (Participants) | 136 | 124
  CFB at Week 33 n=136,124 | 0.036 (0.1996) | 0.055 (0.2595)
  CFB at Week 36 n=129,119: number analyzed (Participants) | 129 | 119
  CFB at Week 36 n=129,119 | 0.061 (0.1767) | 0.054 (0.2881)
  CFB at Week 39 n=133,119: number analyzed (Participants) | 133 | 119
  CFB at Week 39 n=133,119 | 0.037 (0.2015) | 0.071 (0.2816)
  CFB at Week 42 n=124,102: number analyzed (Participants) | 124 | 102
  CFB at Week 42 n=124,102 | 0.044 (0.1794) | 0.063 (0.2680)
  CFB at Week 45 n=124,100: number analyzed (Participants) | 124 | 100
  CFB at Week 45 n=124,100 | 0.035 (0.1961) | 0.065 (0.2584)
  CFB at Week 48 n=111,105: number analyzed (Participants) | 111 | 105
  CFB at Week 48 n=111,105 | 0.056 (0.1870) | 0.081 (0.2603)
  CFB at Week 51 n=103,95: number analyzed (Participants) | 103 | 95
  CFB at Week 51 n=103,95 | 0.026 (0.1682) | 0.067 (0.2840)
  CFB at Week 54 n=104,90: number analyzed (Participants) | 104 | 90
  CFB at Week 54 n=104,90 | 0.043 (0.1703) | 0.054 (0.3086)
  CFB at Week 57 n=109,86: number analyzed (Participants) | 109 | 86
  CFB at Week 57 n=109,86 | 0.037 (0.2012) | 0.049 (0.2979)
  CFB at Week 60 n=94,84: number analyzed (Participants) | 94 | 84
  CFB at Week 60 n=94,84 | 0.022 (0.2119) | 0.069 (0.2819)
  CFB at Week 63 n=94,76: number analyzed (Participants) | 94 | 76
  CFB at Week 63 n=94,76 | 0.034 (0.2056) | 0.082 (0.3043)
  CFB at Week 66 n=89,79: number analyzed (Participants) | 89 | 79
  CFB at Week 66 n=89,79 | 0.026 (0.2011) | 0.071 (0.2996)
  CFB at Week 69 n=93,74: number analyzed (Participants) | 93 | 74
  CFB at Week 69 n=93,74 | 0.052 (0.1805) | 0.061 (0.2964)
  CFB at Week 72 n=87,70: number analyzed (Participants) | 87 | 70
  CFB at Week 72 n=87,70 | 0.032 (0.1890) | 0.057 (0.3176)
  CFB at Week 75 n=78,69: number analyzed (Participants) | 78 | 69
  CFB at Week 75 n=78,69 | 0.021 (0.1797) | 0.080 (0.2966)
  CFB at Week 78 n=77,64: number analyzed (Participants) | 77 | 64
  CFB at Week 78 n=77,64 | 0.027 (0.1979) | 0.056 (0.3064)
  CFB at Week 81 n=73,61: number analyzed (Participants) | 73 | 61
  CFB at Week 81 n=73,61 | 0.035 (0.1844) | 0.042 (0.3529)
  CFB at Week 84 n=63,59: number analyzed (Participants) | 63 | 59
  CFB at Week 84 n=63,59 | 0.056 (0.1923) | 0.064 (0.3125)
  CFB at Week 87 n=44,43: number analyzed (Participants) | 44 | 43
  CFB at Week 87 n=44,43 | 0.049 (0.1894) | 0.057 (0.3474)
  CFB at Week 90 n=37,30: number analyzed (Participants) | 37 | 30
  CFB at Week 90 n=37,30 | 0.050 (0.1610) | 0.039 (0.3502)
  CFB at Week 93 n=24,24: number analyzed (Participants) | 24 | 24
  CFB at Week 93 n=24,24 | 0.082 (0.1861) | 0.074 (0.4112)
  CFB at Week 96 n=19,14: number analyzed (Participants) | 19 | 14
  CFB at Week 96 n=19,14 | 0.071 (0.1604) | 0.018 (0.3986)
  CFB at Week 99 n=15,9: number analyzed (Participants) | 15 | 9
  CFB at Week 99 n=15,9 | 0.116 (0.1755) | 0.099 (0.4211)
  CFB at Week 102 n=8,4: number analyzed (Participants) | 8 | 4
  CFB at Week 102 n=8,4 | 0.144 (0.1730) | -0.002 (0.4701)
  CFB at Week 105 n=5,2: number analyzed (Participants) | 5 | 2
  CFB at Week 105 n=5,2 | 0.073 (0.1476) | -0.232 (0.2489)
  CFB at Week 108 n=1,0: number analyzed (Participants) | 1 | 0
  CFB at Week 108 n=1,0 | 0.121 (NA) — Standard deviation was not calculable due the single data point for the mean value. |
  CFB at Efficacy Follow-up 1 n=9,10: number analyzed (Participants) | 9 | 10
  CFB at Efficacy Follow-up 1 n=9,10 | -0.085 (0.2034) | -0.153 (0.4494)
  CFB at Efficacy Follow-up 2 n=2,4: number analyzed (Participants) | 2 | 4
  CFB at Efficacy Follow-up 2 n=2,4 | -0.031 (0.6781) | -0.195 (0.4873)
  CFB at Efficacy Follow-up 3 n=2,1: number analyzed (Participants) | 2 | 1
  CFB at Efficacy Follow-up 3 n=2,1 | 0.406 (0.4349) | 0.163 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  CFB at Efficacy Follow-up 4 n=0,1: number analyzed (Participants) | 0 | 1
  CFB at Efficacy Follow-up 4 n=0,1 |  | 0.292 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  CFB at CFB at Efficacy Follow-up 5 n=1,0: number analyzed (Participants) | 1 | 0
  CFB at CFB at Efficacy Follow-up 5 n=1,0 | -0.144 (NA) — Standard deviation was not calculable due the single data point for the mean value. |
  CFB at Post-disease Progression (7 days) n=32,24: number analyzed (Participants) | 32 | 24
  CFB at Post-disease Progression (7 days) n=32,24 | -0.126 (0.2115) | -0.048 (0.2844)
  CFB at Post-disease Progression (28 days) n=30,30: number analyzed (Participants) | 30 | 30
  CFB at Post-disease Progression (28 days) n=30,30 | -0.031 (0.2191) | -0.010 (0.2854)

31. Secondary Outcome: Part 2 (Double-blind, Randomized, Placebo-controlled): Change From Baseline in Score as Per the EuroQol 5 Dimension 5 Level (EQ-5D-5L) Questionnaire - Visual Analog Scale (VAS)
Description: The EQ-5D-5L is a standardized questionnaire used to assess health-related quality of life, and it includes a Visual Analog Scale (VAS). The VAS score is obtained by asking the individual to rate their current health status on a scale from 0 to 100, where 0 represents the worst possible health state and 100 represents the best possible health state.
  The change from baseline in EQ-5D-5L VAS score was calculated. A positive change from baseline indicates improvement in the health status. CFB = change from baseline
Time Frame: as for outcome 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 320 | 323
score on a scale
  CFB at Week 3 n=254,249: number analyzed (Participants) | 254 | 249
  CFB at Week 3 n=254,249 | 0.1 (16.51) | 3.2 (18.35)
  CFB at Week 6 n=236,230: number analyzed (Participants) | 236 | 230
  CFB at Week 6 n=236,230 | 1.3 (16.04) | 2.6 (18.18)
  CFB at Week 9 n=220,219: number analyzed (Participants) | 220 | 219
  CFB at Week 9 n=220,219 | 1.4 (15.23) | 2.5 (17.22)
  CFB at Week 12 n=192,214: number analyzed (Participants) | 192 | 214
  CFB at Week 12 n=192,214 | 0.0 (18.28) | 3.3 (16.78)
  CFB at Week 15 n=194,196: number analyzed (Participants) | 194 | 196
  CFB at Week 15 n=194,196 | 0.8 (17.41) | 2.7 (18.72)
  CFB at Week 18 n=187,198: number analyzed (Participants) | 187 | 198
  CFB at Week 18 n=187,198 | 0.4 (16.76) | 4.4 (17.66)
  CFB at Week 21 n=173,176: number analyzed (Participants) | 173 | 176
  CFB at Week 21 n=173,176 | 0.0 (16.92) | 2.3 (18.49)
  CFB at Week 24 n=161,164: number analyzed (Participants) | 161 | 164
  CFB at Week 24 n=161,164 | 0.4 (17.15) | 2.3 (19.40)
  CFB at Week 27 n=158,155: number analyzed (Participants) | 158 | 155
  CFB at Week 27 n=158,155 | 0.1 (16.38) | 2.8 (17.65)
  CFB at Week 30 n=141,145: number analyzed (Participants) | 141 | 145
  CFB at Week 30 n=141,145 | 0.7 (16.45) | 2.5 (19.08)
  CFB at Week 33 n=137,124: number analyzed (Participants) | 137 | 124
  CFB at Week 33 n=137,124 | 0.8 (14.50) | 4.1 (17.00)
  CFB at Week 36 n=130,119: number analyzed (Participants) | 130 | 119
  CFB at Week 36 n=130,119 | 2.3 (14.79) | 4.8 (16.73)
  CFB at Week 39 n=134,119: number analyzed (Participants) | 134 | 119
  CFB at Week 39 n=134,119 | 2.2 (15.25) | 4.6 (16.68)
  CFB at Week 42 n=125,103: number analyzed (Participants) | 125 | 103
  CFB at Week 42 n=125,103 | 1.5 (15.15) | 4.7 (17.17)
  CFB at Week 45 n=125,100: number analyzed (Participants) | 125 | 100
  CFB at Week 45 n=125,100 | 1.2 (16.15) | 5.0 (14.75)
  CFB at Week 48 n=112,105: number analyzed (Participants) | 112 | 105
  CFB at Week 48 n=112,105 | 0.9 (16.62) | 3.9 (17.29)
  CFB at Week 51 n=104,95: number analyzed (Participants) | 104 | 95
  CFB at Week 51 n=104,95 | 0.8 (15.94) | 2.8 (17.07)
  CFB at Week 54 n=104,90: number analyzed (Participants) | 104 | 90
  CFB at Week 54 n=104,90 | 0.5 (14.43) | 4.2 (17.50)
  CFB at Week 57 n=110,86: number analyzed (Participants) | 110 | 86
  CFB at Week 57 n=110,86 | 0.2 (16.63) | 2.1 (19.12)
  CFB at Week 60 n=95,84: number analyzed (Participants) | 95 | 84
  CFB at Week 60 n=95,84 | -1.4 (16.49) | 2.8 (17.46)
  CFB at Week 63 n=95,76: number analyzed (Participants) | 95 | 76
  CFB at Week 63 n=95,76 | 0.0 (17.35) | 3.0 (20.02)
  CFB at Week 66 n=90,79: number analyzed (Participants) | 90 | 79
  CFB at Week 66 n=90,79 | 1.0 (15.49) | 4.6 (19.36)
  CFB at Week 69 n=94,74: number analyzed (Participants) | 94 | 74
  CFB at Week 69 n=94,74 | 1.9 (15.48) | 5.6 (18.30)
  CFB at Week 72 n=88,70: number analyzed (Participants) | 88 | 70
  CFB at Week 72 n=88,70 | 0.4 (15.30) | 3.6 (19.21)
  CFB at Week 75 n=79,69: number analyzed (Participants) | 79 | 69
  CFB at Week 75 n=79,69 | -0.1 (15.96) | 5.1 (19.12)
  CFB at Week 78 n=78,64: number analyzed (Participants) | 78 | 64
  CFB at Week 78 n=78,64 | 0.1 (17.65) | 5.1 (19.34)
  CFB at Week 81 n=73,61: number analyzed (Participants) | 73 | 61
  CFB at Week 81 n=73,61 | 0.2 (16.10) | 3.1 (19.38)
  CFB at Week 84 n=64,59: number analyzed (Participants) | 64 | 59
  CFB at Week 84 n=64,59 | 2.0 (16.33) | 2.0 (19.05)
  CFB at Week 87 n=44,43: number analyzed (Participants) | 44 | 43
  CFB at Week 87 n=44,43 | 0.6 (17.07) | 1.7 (18.35)
  CFB at Week 90 n=37,30: number analyzed (Participants) | 37 | 30
  CFB at Week 90 n=37,30 | -1.9 (17.04) | 2.6 (18.13)
  CFB at Week 93 n=24,24: number analyzed (Participants) | 24 | 24
  CFB at Week 93 n=24,24 | 1.9 (16.06) | 0.7 (16.75)
  CFB at Week 96 n=19,14: number analyzed (Participants) | 19 | 14
  CFB at Week 96 n=19,14 | 2.9 (15.01) | 4.8 (16.28)
  CFB at Week 99 n=15,9: number analyzed (Participants) | 15 | 9
  CFB at Week 99 n=15,9 | -1.2 (12.09) | 5.9 (19.51)
  CFB at Week 102 n=8,4: number analyzed (Participants) | 8 | 4
  CFB at Week 102 n=8,4 | 5.3 (14.98) | 0.5 (21.63)
  CFB at Week 105 n=5,2: number analyzed (Participants) | 5 | 2
  CFB at Week 105 n=5,2 | 7.2 (19.49) | -15.5 (7.78)
  CFB at Week 108 n=1,0: number analyzed (Participants) | 1 | 0
  CFB at Week 108 n=1,0 | 3.0 (NA) — Standard deviation was not calculable due the single data point for the mean value. |
  CFB at Efficacy Follow-up 1 n=9,10: number analyzed (Participants) | 9 | 10
  CFB at Efficacy Follow-up 1 n=9,10 | -1.6 (17.67) | -9.8 (27.85)
  CFB at Efficacy Follow-up 2 n=2,4: number analyzed (Participants) | 2 | 4
  CFB at Efficacy Follow-up 2 n=2,4 | 8.5 (9.19) | -5.3 (17.23)
  CFB at Efficacy Follow-up 3 n=2,1: number analyzed (Participants) | 2 | 1
  CFB at Efficacy Follow-up 3 n=2,1 | 12.5 (19.09) | 5.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  CFB at Efficacy Follow-up 4 n=0,1: number analyzed (Participants) | 0 | 1
  CFB at Efficacy Follow-up 4 n=0,1 |  | 21.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  CFB at CFB at Efficacy Follow-up 5 n=1,0: number analyzed (Participants) | 1 | 0
  CFB at CFB at Efficacy Follow-up 5 n=1,0 | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value. |
  CFB at Post-disease Progression (7 days) n=32,24: number analyzed (Participants) | 32 | 24
  CFB at Post-disease Progression (7 days) n=32,24 | -10.4 (18.36) | -4.6 (21.40)
  CFB at Post-disease Progression (28 days) n=30,30: number analyzed (Participants) | 30 | 30
  CFB at Post-disease Progression (28 days) n=30,30 | -0.1 (19.14) | -1.4 (22.92)

32. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths due to any cause were collected from first dose of study medication to 30 days after the last dose of study treatment. Post-treatment survival follow-up deaths were collected from Day 31 after last dose of study medication to the data cut-off date.
Time Frame: On-treatment deaths: Up to approximately 29 months in Part 1 or approximately 25 months in Part 2. Post-treatment survival follow-up deaths: Up to an additional 130 days.
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned and who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A | Part 1: Cohort B | Part 1: Cohort C | Part 2: Canakinumab+Pembro+CTx | Part 2: Placebo+Pembro+CTx
Number analyzed (Participants) | 10 | 11 | 9 | 320 | 323
Participants
  Pre-treatment deaths | 0 | 0 | 0 | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 10 | 11 | 9 | 320 | 322
  On-treatment deaths | 4 | 1 | 4 | 97 | 102
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 6 | 10 | 5 | 223 | 220
  Post-treatment survival follow-up deaths | 2 | 5 | 3 | 50 | 57
  All deaths | 6 | 6 | 7 | 147 | 159

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 32 months.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients that entered the post-treatment survival follow-up period. All-cause Mortality was assessed on the Full analysis set (FAS). SAEs and AEs were assessed on the Safety Set (participants who received at least one dose of the study treatment).
Groups:
- Part 1: Cohort A (On-treatment); Part 1: Cohort B (On-treatment); Part 1: Cohort C (On-treatment); Part 2: Canakinumab+Pembro+CTx (On-treatment); Part 2: Placebo+Pembro+CTx (On-treatment): AEs during the on-treatment period (up to 30 days post-treatment)
- Part 1: Cohort A (Post-treatment Survival Follow-up); Part 1: Cohort B (Post-treatment Survival Follow-up); Part 1: Cohort C (Post-treatment Survival Follow-up); Part 2: Canakinumab+Pembro+CTx (Post-treatment Survival Follow-up); Part 2: Placebo+Pembro+CTx (Post-treatment Survival Follow-up): Deaths collected in the post-treatment survival follow-up period (starting from Day 31 post-treatment). No AEs were collected during this period.
Arm/Group | Part 1: Cohort A (On-treatment) | Part 1: Cohort B (On-treatment) | Part 1: Cohort C (On-treatment) | Part 2: Canakinumab+Pembro+CTx (On-treatment) | Part 2: Placebo+Pembro+CTx (On-treatment) | Part 1: Cohort A (Post-treatment Survival Follow-up) | Part 1: Cohort B (Post-treatment Survival Follow-up) | Part 1: Cohort C (Post-treatment Survival Follow-up) | Part 2: Canakinumab+Pembro+CTx (Post-treatment Survival Follow-up) | Part 2: Placebo+Pembro+CTx (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 4/10 | 1/11 | 4/9 | 97/320 | 102/323 | 2/6 | 5/10 | 3/5 | 50/223 | 57/220
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/11 | 4/9 | 174/320 | 167/322 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11 | 9/9 | 309/320 | 310/322 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort A (On-treatment) (N=10) | Part 1: Cohort B (On-treatment) (N=11) | Part 1: Cohort C (On-treatment) (N=9) | Part 2: Canakinumab+Pembro+CTx (On-treatment) (N=320) | Part 2: Placebo+Pembro+CTx (On-treatment) (N=322) | Part 1: Cohort A (Post-treatment Survival Follow-up) (N=0) | Part 1: Cohort B (Post-treatment Survival Follow-up) (N=0) | Part 1: Cohort C (Post-treatment Survival Follow-up) (N=0) | Part 2: Canakinumab+Pembro+CTx (Post-treatment Survival Follow-up) (N=0) | Part 2: Placebo+Pembro+CTx (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 10 | 11 | NA | NA | NA | NA | NA
Bicytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 10 | 8 | NA | NA | NA | NA | NA
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Immune-mediated cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 7 | 8 | NA | NA | NA | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2 | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4 | 1 | NA | NA | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 2 | 3 | NA | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 2 | 3 | NA | NA | NA | NA | NA
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 3 | 2 | NA | NA | NA | NA | NA
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 4 | 1 | NA | NA | NA | NA | NA
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 4 | 1 | NA | NA | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Adrenal disorder (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 1 | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 7 | 10 | NA | NA | NA | NA | NA
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 3 | NA | NA | NA | NA | NA
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 5 | 2 | NA | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 4 | NA | NA | NA | NA | NA
Chest pain (General disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 0 | 2 | 3 | NA | NA | NA | NA | NA
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Implant site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Performance status decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 0 | 0 | 1 | 12 | 8 | NA | NA | NA | NA | NA
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 4 | NA | NA | NA | NA | NA
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 5 | 6 | NA | NA | NA | NA | NA
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | NA | NA | NA | NA | NA
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Empyema (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Gastrointestinal protozoal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 4 | 1 | NA | NA | NA | NA | NA
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Nosocomial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 32 | 25 | NA | NA | NA | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | NA | NA | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 4 | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 6 | 10 | NA | NA | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 0 | 0 | 5 | 3 | NA | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 3 | NA | NA | NA | NA | NA
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 4 | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Cortisol decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 6 | 1 | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 0 | 6 | 0 | NA | NA | NA | NA | NA
Transaminases increased (Investigations) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 2 | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 4 | NA | NA | NA | NA | NA
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 5 | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 5 | NA | NA | NA | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 3 | NA | NA | NA | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 16 | 13 | NA | NA | NA | NA | NA
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 6 | NA | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 9 | 8 | NA | NA | NA | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 9 | 6 | NA | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 8 | 6 | NA | NA | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4 | NA | NA | NA | NA | NA
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort A (On-treatment) (N=10) | Part 1: Cohort B (On-treatment) (N=11) | Part 1: Cohort C (On-treatment) (N=9) | Part 2: Canakinumab+Pembro+CTx (On-treatment) (N=320) | Part 2: Placebo+Pembro+CTx (On-treatment) (N=322) | Part 1: Cohort A (Post-treatment Survival Follow-up) (N=0) | Part 1: Cohort B (Post-treatment Survival Follow-up) (N=0) | Part 1: Cohort C (Post-treatment Survival Follow-up) (N=0) | Part 2: Canakinumab+Pembro+CTx (Post-treatment Survival Follow-up) (N=0) | Part 2: Placebo+Pembro+CTx (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 3 | 153 | 148 | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 26 | 15 | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 124 | 78 | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 58 | 42 | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 3 | 6 | NA | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 1 | 2 | NA | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 2 | 2 | NA | NA | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 2 | 3 | 1 | NA | NA | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 5 | 3 | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 2 | 19 | 14 | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 1 | 2 | 1 | 31 | 28 | NA | NA | NA | NA | NA
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Dry eye (Eye disorders) | 1 | 1 | 0 | 4 | 7 | NA | NA | NA | NA | NA
Endocrine ophthalmopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Lacrimation increased (Eye disorders) | 0 | 3 | 0 | 9 | 7 | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1 | 4 | NA | NA | NA | NA | NA
Visual impairment (Eye disorders) | 1 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Xerophthalmia (Eye disorders) | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 5 | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1 | 14 | 19 | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 10 | 5 | NA | NA | NA | NA | NA
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 6 | 3 | 2 | 84 | 81 | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 61 | 66 | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 10 | 5 | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 9 | 9 | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 7 | 9 | NA | NA | NA | NA | NA
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 3 | 5 | 5 | 115 | 124 | NA | NA | NA | NA | NA
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 3 | NA | NA | NA | NA | NA
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 11 | 17 | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 | 5 | 2 | 54 | 51 | NA | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 3 | 1 | 93 | 87 | NA | NA | NA | NA | NA
Chest discomfort (General disorders) | 0 | 1 | 0 | 4 | 5 | NA | NA | NA | NA | NA
Chest pain (General disorders) | 1 | 2 | 1 | 18 | 18 | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 1 | 0 | 4 | 1 | NA | NA | NA | NA | NA
Effusion (General disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Fatigue (General disorders) | 2 | 5 | 3 | 59 | 68 | NA | NA | NA | NA | NA
Generalised oedema (General disorders) | 0 | 1 | 0 | 7 | 1 | NA | NA | NA | NA | NA
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Injection site reaction (General disorders) | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Malaise (General disorders) | 1 | 1 | 1 | 8 | 6 | NA | NA | NA | NA | NA
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 17 | 17 | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 3 | 5 | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 1 | 1 | 1 | 35 | 42 | NA | NA | NA | NA | NA
Pain (General disorders) | 0 | 1 | 0 | 9 | 8 | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 1 | 0 | 4 | 3 | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 2 | 2 | 1 | 44 | 65 | NA | NA | NA | NA | NA
Swelling (General disorders) | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Swelling face (General disorders) | 0 | 1 | 0 | 3 | 1 | NA | NA | NA | NA | NA
Allergic reaction to excipient (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Borrelia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Candida infection (Infections and infestations) | 1 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 10 | 13 | NA | NA | NA | NA | NA
Eye infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 5 | 7 | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 8 | 6 | NA | NA | NA | NA | NA
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 3 | 2 | NA | NA | NA | NA | NA
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 3 | 3 | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 26 | 16 | NA | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | NA | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 1 | 18 | 15 | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 19 | 20 | NA | NA | NA | NA | NA
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Viral rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 8 | 4 | NA | NA | NA | NA | NA
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 76 | 50 | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 0 | 0 | 32 | 39 | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 62 | 47 | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 25 | 22 | NA | NA | NA | NA | NA
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 6 | 2 | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 28 | 42 | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 49 | 37 | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 2 | 1 | 0 | 19 | 31 | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 27 | 14 | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 3 | 3 | 1 | 79 | 58 | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 2 | 1 | 0 | 50 | 32 | NA | NA | NA | NA | NA
SARS-CoV-2 test negative (Investigations) | 0 | 1 | 0 | 36 | 42 | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 0 | 2 | 0 | 31 | 30 | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 2 | 2 | 0 | 63 | 43 | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 1 | 91 | 79 | NA | NA | NA | NA | NA
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 7 | 6 | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 24 | 26 | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 20 | 16 | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 33 | 32 | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 25 | 34 | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 24 | 18 | NA | NA | NA | NA | NA
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 49 | 56 | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 26 | 32 | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 8 | 7 | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 5 | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 10 | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 13 | 11 | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 25 | 28 | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 6 | 9 | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 22 | 22 | NA | NA | NA | NA | NA
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 3 | NA | NA | NA | NA | NA
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 23 | 21 | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 15 | 16 | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 1 | 0 | 21 | 33 | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 4 | 9 | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 4 | 22 | 18 | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 2 | 3 | 24 | 20 | NA | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 6 | 6 | NA | NA | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 5 | 1 | NA | NA | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | NA | NA | NA | NA | NA
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 11 | 11 | NA | NA | NA | NA | NA
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 29 | 31 | NA | NA | NA | NA | NA
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 5 | 5 | NA | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 5 | 7 | NA | NA | NA | NA | NA
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 54 | 51 | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 59 | 61 | NA | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 9 | 11 | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 16 | 22 | NA | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4 | 8 | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 10 | 5 | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 16 | 21 | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 8 | 5 | NA | NA | NA | NA | NA
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 29 | 31 | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 15 | 14 | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 7 | 1 | NA | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5 | 9 | NA | NA | NA | NA | NA
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 48 | 43 | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 5 | 2 | 51 | 61 | NA | NA | NA | NA | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 10 | 10 | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 5 | NA | NA | NA | NA | NA
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Hot flush (Vascular disorders) | 0 | 0 | 1 | 3 | 4 | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 2 | 1 | 24 | 22 | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | 0 | 13 | 6 | NA | NA | NA | NA | NA
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03631199/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03631199/SAP_001.pdf